CLINICAL TRIAL: NCT06540521
Title: Intracardiac Electrical Characteristics of LBBAP
Brief Title: Bolt CSP-M Holter Study
Status: Recruiting | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT24030
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Bradycardia
Keywords: LBBAP; LBBP; LVSP
MeSH Terms: conditions — Heart Failure; Bradycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to investigate the cardiac electrical characteristics in different pacing outputs and body positions in LBB area pacing (LBBAP), from which the findings may help to develop and support data validation of a novel algorithm for LBB capture determination for LBBAP.

DETAILED DESCRIPTION:
Among LBB area pacing (LBBAP), it has been reported that left ventricular (LV) septal pacing (LVSP), which refers to a pacing approach that only captures the LV septal myocardium, produces homogeneous electrical propagation in the septum and leads to delayed LV lateral wall activation. Although large randomized trials are lacking, small observational studies have shown more preserved physiological ventricular depolarization, or superior electrical and mechanical synchrony of the LBB capture over LVSP.

During the implantation of a device, the most commonly used method to distinguish LVSP from the LBB capture is to pace with different pacing outputs. A transition will be found in the ECG morphology with changes in the LV activation time if the pacing capture threshold (PCT) of the local myocardium is different from that of the LBB (i.e., LBB-PCT), indicating a transition between capturing the LBB and LVSP without any LBB capture. So far, there is no systematic investigation on the EGM characteristics or correlation between ECG and EGM characteristics at different conduction system capture status. Findings from this study will help to better characterize EGM characteristics and to develop an optimal LBBAP modality to differentiate LBB capture.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >=18 years
* Patients who are willing to provide Informed Consent
* Patients who have received LBBAP therapy >= 1 month for 1 to 4 months (including 1 and 4 month)
* Patients implanted with a single/dual-chamber pacemaker or a CRT-P with LBBAP lead connected to RV port
* Implanted device can provide at least 3-channel real-time intracardiac electrogram

Exclusion Criteria:

* Patients who are pregnant or have a plan for pregnancy during the study
* Patients who have medical conditions that would limit study participation
* Patients who were already enrolled in clinical trial(s) which would impact study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study selected two study site in China. One is a Tertiary A hospital in Shanghai, and another is a cardiovascular specialty hospital in Zhejiang Province. Both the two sites locate in the south east of China. This study will enroll 70 subjects who meet all the inclusion and exclusion criteria from the patients who have received LBBAP therapies from the two hospitals.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Intracardiac electrical characteristics in different pacing outputs. | received LBBAP therapy >= 1 month for 1 to 4 months (including 1 and 4 month); and an optional follow-up 6 month after the enrollment
  12-lead ECG and LBBAP EGM characteristics and duration in different pacing outputs.

SECONDARY OUTCOMES:
Intracardiac electrical characteristics under different body position. | received LBBAP therapy >= 1 month for 1 to 4 months (including 1 and 4 month); and an optional follow-up 6 month after the enrollment
  12-lead ECG and LBBAP EGM characteristics and duration under different body positions.
The correlation between LBB capture status and LBBAP EGM characteristics | received LBBAP therapy >= 1 month for 1 to 4 months (including 1 and 4 month); and an optional follow-up 6 month after the enrollment
  ECG and EGM characteristics in different LBB capture status

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Greentown Cardiovascular Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang W, Su L, Wu S, Xu L, Xiao F, Zhou X, Ellenbogen KA. A Novel Pacing Strategy With Low and Stable Output: Pacing the Left Bundle Branch Immediately Beyond the Conduction Block. Can J Cardiol. 2017 Dec;33(12):1736.e1-1736.e3. doi: 10.1016/j.cjca.2017.09.013. Epub 2017 Sep 22. PMID 29173611
- [Background] Chen X, Qian Z, Zou F, Wang Y, Zhang X, Qiu Y, Hou X, Zhou X, Vijayaraman P, Zou J. Differentiating left bundle branch pacing and left ventricular septal pacing: An algorithm based on intracardiac electrophysiology. J Cardiovasc Electrophysiol. 2022 Mar;33(3):448-457. doi: 10.1111/jce.15350. Epub 2022 Jan 12. PMID 34978368
- [Background] Zhou Y, Wang J, Wei Y, Zhang W, Yang Y, Rui S, Ju C. Left ventricular septal pacing versus left bundle branch pacing in the treatment of atrioventricular block. Ann Noninvasive Electrocardiol. 2022 May;27(3):e12944. doi: 10.1111/anec.12944. Epub 2022 Mar 10. PMID 35267228
- [Background] Wu S, Chen X, Wang S, Xu L, Xiao F, Huang Z, Zheng R, Jiang L, Vijayaraman P, Sharma PS, Su L, Huang W. Evaluation of the Criteria to Distinguish Left Bundle Branch Pacing From Left Ventricular Septal Pacing. JACC Clin Electrophysiol. 2021 Sep;7(9):1166-1177. doi: 10.1016/j.jacep.2021.02.018. Epub 2021 Apr 28. PMID 33933414